CLINICAL TRIAL: NCT00276913
Title: A Phase I Study of STA-5312 Administered Weekly in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Study of STA-5312 in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5312-02
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Advanced or Metastatic Solid Tumors

INTERVENTIONS:
Drug: STA-5312

SUMMARY:
Primary Objectives:

* To determine the safety, toxicity and the maximum tolerated dose (MTD) of intravenous STA-5312 when administered weekly (3 of 4 weeks) to subjects with advanced or metastatic solid tumors.
* To determine the pharmacokinetics of STA-5312.

Secondary Objective:

• To assess antitumor activity of STA-5312 administration.

DETAILED DESCRIPTION:
This is a Phase I open-label, dose-escalation safety study in subjects with refractory non hematologic malignancies. STA-5312 will be administered intravenously. Administration is anticipated to take 1 hour, although infusion time may be extended when appropriate with large infusion volumes. A treatment cycle is 4 weeks with a weekly infusion of STA 5312 for the first 3 weeks of each 4 week cycle. The planned treatment schedule is 2 cycles of STA-5312 treatment (8 weeks). Decisions regarding dose escalation and DLT determination will be made based on observations during the first cycle of therapy. Subjects who tolerate treatment may be eligible to continue receiving additional cycles of STA 5312 per the investigator's medical judgment. Evaluation of antitumor response will be performed after every 2 cycles of STA 5312 administration.

The initial dose level of STA 5312 will be 6 mg/m2. The starting dose level was chosen based on preclinical animal studies that used alternate day dosing x 3/week on alternate weeks. The dose level of 6 mg/m2 represents less than 1/10 the weekly dose (3 mg/m2 x 3) that demonstrated severe toxicity. Subsequent dose escalations will follow an accelerated titration design once the 8 mg/m2 cohort is completed No fewer than 3 patients will be enrolled at each dose level. Once a DLT is observed the cohort will be expanded to at least six subjects. If one-third of at least 6 subjects treated at a dose level experience a DLT, dose escalation will terminate. The dose below this will be considered the MTD and will be expanded to at least 12 subjects to collect additional safety and pharmacokinetic data. No intrasubject dose escalations will occur.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged at least 18 years with histologically-confirmed non hematological malignancy that is metastatic or unresectable and for which no standard therapy exists.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2.
* Peripheral neuropathy less than Grade 2 on National Cancer Institute Common Toxicity Criteria (NCI CTC) version 3 adverse event scale.
* Subjects must have acceptable organ and marrow function during the Screening Period as defined below. (Note: Subjects must meet these criteria at each pre-dose visit to receive additional doses of STA-5312).

  * Absolute neutrophil count (ANC) greater than 1500 cells/µL
  * Platelets greater than 100,000/µL
  * Total bilirubin must be <1.5 times ULN
  * Aspartate transaminase (AST) ≤3 times ULN or less than 5 times the ULN in subjects with liver metastases
  * Alanine transaminase (ALT) ≤3 times ULN or less than 5 times the ULN in subjects with liver metastases
  * Adequate renal function (serum creatinine <2.0 mg/dL).
* Electrocardiogram (ECG) without evidence of clinically significant ventricular arrhythmias or active ischemia as determined by the investigator.
* Documented cardiac ejection fraction greater than 50% obtained within 30 days of administration of the first dose.
* The effects of STA-5312 on the developing human fetus are unknown. Therefore, women of childbearing potential (defined as women over 50 years of age or history of amenorrhea for <12 months prior to study entry) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a female subject become pregnant or suspect she is pregnant while participating in this study, she should inform the treating physician immediately.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Women who are pregnant or breast-feeding.
* Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Subjects with previous high-dose chemotherapy with autologous allogeneic hematopoietic stem cell transplantation.
* Subjects with primary brain tumors or active brain metastases are excluded. Subjects with previously treated brain metastases who are not receiving corticosteroids or anticonvulsants are eligible.
* History of stroke within 6 months of treatment or other significant neurological limitations.
* Use of any investigational agents within 4 weeks of study enrollment.
* History of severe allergic reactions to excipients (e.g. Tween 80/polysorbate 80), including severe hypersensitivity reactions defined as greater than Grade 3 based on NCI CTC version 3.
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-06

CONTACTS AND LOCATIONS:
Locations (1):
- Steven Limentani, MD, Charlotte, North Carolina, United States